CLINICAL TRIAL: NCT00324714
Title: A Randomised, Double-Blind Trial to Assess the Effects on Bone Mineral Density and Bone Biomarkers of Anastrozole When Used to Prevent Breast Cancer in Postmenopausal Women
Brief Title: Risedronate in Improving Bone Mineral Density and Bone Health in Postmenopausal Women With Ductal Carcinoma In Situ Enrolled in Clinical Trial CRUK-IBIS-II-DCIS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000474949; IBCSG-31-03-PBS; EUDRACT-2004-003991-12
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Risedronic Acid

INTERVENTIONS:
Drug: risedronate sodium
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Bisphosphonates, such as risedronate, may help improve bone health and prevent osteoporosis in postmenopausal women. It is not yet known whether risedronate is effective in improving bone mineral density and bone health in women with ductal carcinoma in situ.

PURPOSE: This randomized phase III trial is studying risedronate to see how well it works compared to a placebo in improving bone mineral density and bone health in postmenopausal women with ductal carcinoma in situ enrolled in clinical trial CRUK-IBIS-II-DCIS (CRUK: Cancer Research UK) (DCIS: Ductal carcinoma in situ).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the changes in bone of the spine and femur in postmenopausal women with ductal carcinoma in situ treated with anastrozole vs placebo on protocol CRUK-IBIS-II-DCIS.
* Determine the effect of bisphosphonate treatment on bone mineral density and bone metabolism in patients who are receiving anastrozole on protocol CRUK-IBIS-II-DCIS and are osteoporotic or moderately to severely osteopenic at baseline.

Secondary

* Correlate changes in levels of biochemical markers of bone metabolism with longer-term changes in bone mineral density, as measured by dual-energy x-ray absorptiometry (DXA).

OUTLINE: This is a multicenter, partially randomized, double-blind study. Patients are stratified according to bone mineral density (T-score) measurements (≥ -1.5 vs -2.5 to < -1.5 vs -4.0 to < -2.5 or ≤ 2 low-trauma vertebral fractures). Patients in stratum I are further stratified according to calcium and cholecalciferol (vitamin D) supplementation (yes vs no) and use of risedronate on this study (yes vs no). Patients in stratum II are further stratified according to randomized treatment on protocol CRUK-IBIS-II-DCIS (yes vs no).

* Stratum I (T-score ≥ -1.5): Patients undergo dual-energy x-ray absorptiometry (DXA) scanning at baseline and then at 1, 3, 5, and 7 years. Patients who develop osteoporosis (T-score < -2.5) are removed from the study and receive open-label bisphosphonates.
* Stratum II (T-score -2.5 to < -1.5 [moderate to severe osteopenia]): Patients undergo DXA scanning as in stratum I. Patients are also randomized (double-blind) to 1 of 2 treatment arms.

  * Arm I: Patients receive oral risedronate once a week for 5 years.
  * Arm II: Patients receive oral placebo once a week for 5 years. Patients in either arm who develop osteoporosis AND a drop in T-score of more than 1 unit are removed from the study and receive open-label bisphosphonates.
* Stratum III (T-score -4.0 to < -2.5 OR ≤ 2 low trauma vertebral fractures [osteoporosis]): Patients undergo DXA scanning as in stratum I. Patients also receive oral risedronate (or their current bisphosphonate) once a week for 5 years.

Blood samples for correlative studies (e.g., bone biomarkers, serum estradiol) are collected at baseline and at 6 and 12 months.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ductal carcinoma in situ within the past 6 months

  * Locally excised with tumor-free margins at least 1 mm
* Currently enrolled in protocol CRUK-IBIS-II-DCIS AND randomized to receive either anastrozole or placebo
* No T-score < -4.0 and/or > 2 low trauma vertebral fractures by dual-energy x-ray absorptiometry (DXA)
* Hormone receptor status: Estrogen or progesterone receptor positive tumor

PATIENT CHARACTERISTICS:

* Female patient
* Postmenopausal
* No prior bilateral hip fracture or bilateral hip prostheses
* No concurrent metabolic bone disease, including any of the following:

  * Paget's disease
  * Osteogenesis imperfecta
  * Disorders of calcium or mineral metabolism
  * Renal calculus
  * Malabsorption
  * Hypercalcemia or hypocalcemia
  * Hyperparathyroidism or hypoparathyroidism
  * Hyperthyroidism or hypothyroidism

    * Patients on stable replacement therapy are allowed provided they are euthyroid

PRIOR CONCURRENT THERAPY:

* More than 12 months since prior medication affecting bone metabolism, including any of the following:

  * Estrogen
  * Any bisphosphonate
  * Parathyroid hormone
  * Calcitonin
  * Oral or systemic glucocorticoids

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-02

PRIMARY OUTCOMES:
Spine and femur bone change comparison
Effects of bisphosphonate on bone mineral density and bone metabolism in patients who were osteoporotic or moderately severe osteopenic at baseline

SECONDARY OUTCOMES:
Correlation of changes in levels of biochemical markers of bone metabolism with longer-term changes in bone mineral density as measured by dual-energy x-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina S. Buser, MD, Principal Investigator — Oncocare Sonnenhof-Klinik Engeriedspital
Locations (2):
- Switzerland (2):
  - Inselspital Bern, Bern
  - Oncocare Sonnenhof-Klinik Engeriedspital, Bern

REFERENCES:
- [Result] Singh S, Cuzick J, Edwards R, et al.: Effect of anastrozole on bone mineral density after one year of treatment: results from bone sub-study of the International Breast Cancer Intervention Study (IBIS-II). [Abstract] Breast Cancer Res Treat 106 (1): A-28, S9, 2007.
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716